CLINICAL TRIAL: NCT02334852
Title: Registry of Atrial Fibrillation and Embolic Risk in Mexico
Acronym: CARMEN-AF
Status: Completed | Type: Observational
Sponsor: Registro de Fibrilación Auricular y Riesgo Embólico en México (Other)
Collaborators: Bayer (Industry); Boehringer Ingelheim (Industry); Bristol-Myers Squibb (Industry); Pfizer (Industry); Medicaweb, S.A.C.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CARMEN
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The AF is the most common arrhythmia in clinical practice affecting 1-2% of the general population. It is the most common cause of cerebrovascular events (CVE), responsible for 25% of all ischemic strokes and 50% of cardioembolic strokes.

The CARMEN-AF registry is planned to be the first registry of non-valvular AF in Mexico with national representation, planning and specific objectives for publications. Follow-up period of two years is planned.

DETAILED DESCRIPTION:
The CARMEN-AF registry intends to achieve a national sample of non-valvular AF in male and female patients older than 18 years through the participation of every state of Mexico. Thus, a wide geographical distribution will allow comparing health care quality between different geographical areas in which the patients are attended (Northwest, North, Center, Mexico City, East and Southeast).

Besides, to guarantee this national representation, the principle health institutions are planned to participate, the public and the private ones.

Primary objectives:

To know the current state of thromboprophylaxis in non-valvular Atrial Fibrillation (AF) in Mexico.

To evaluate the therapeutic behavior according to the Clinical Practice Guidelines (CPG) at baseline and one year follow-up, with an educational strategy to increase the adherence.

Secondary objectives:

To identify the characteristics of oral anticoagulants current use in Mexico.

To analyze the efficiency of anticoagulation with vitamin K antagonists and the new oral anticoagulants, at baseline and one year follow-up.

Descriptive statistics:

For each group of variables the following descriptive statistics will be obtained:

In continuous variables: mean, standard deviation (SD), standard error, confidence interval (CI) 95%, minimum, percentile 25, median, percentile75, maximum, n and number of lost data.

In categorical variables: % from total column, n in each category. Lost data will be treated as a new category.

Ethical aspects:

Every investigator should fulfil the study according with the principles of the Helsinki declaration.

Copies of the Helsinki Declaration and its subsequent amendments will be provided under specific request or can be obtained through the World Medical Association website (http://www.wma.net/en/30publications /10policies/b3/index.html).

The study should be developed in accordance with the protocol and the procedures that ensure the standards of Good Clinical Practice (GCP) compliance (1996).

The study will be conducted in accordance with the guidelines for Good Epidemiological Practice.

Risk-benefit assessment for the research subjects:

Patients included in the study are not subject to experimental considerations.

Information sheet and informed consent form:

As this study represents a longitudinal observational registry that does not imply therapeutic change, no informed consent form is contemplated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented diagnosis of AF in the last six months by 12-lead electrocardiogram, rhythm strip, or Holter monitoring, pacemaker minimum 30 seconds (with or without treatment and regardless of rhythm during enrollment)
* Patients presenting AF (diagnosed by standard ECG or Holter monitoring) at baseline
* Patients should be eligible for treatment with oral anticoagulant thromboprophylaxis
* Patients with at least 1 risk factor for thromboembolism (CVE or outside the CNS) according to CHA2DS2VASc

Exclusion Criteria:

* AF of transient causes (thyrotoxicosis, alcohol intoxication, myocardial infarction (MI) acute phase, pericarditis, myocarditis, electrocution, pulmonary embolism or other lung disease, electrolyte or metabolic disorder,etc).
* AF onset in immediate postoperative or 3 months in cardiac surgery
* Terminal illness
* Mental Inability to take anticoagulants
* Inability to fulfill the follow-up visits
* Programming for ablation of pulmonary veins
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented diagnosis of AF in the last six months
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Oral anticoagulation | One year
  To analyze quality of anticoagulation with vitamin K antagonists at baseline (control) and one year.

CONTACTS AND LOCATIONS:
Overall Officials: Manlio F Marquez-Murillo, MD, Principal Investigator — Instituto Nacional de Cardiología

REFERENCES:
- [Derived] Marquez MF, Banos-Gonzalez MA, Guevara-Valdivia ME, Vazquez-Acosta J, de Los Rios Ibarra MO, Aguilar-Linares JA, Jimenez-Cruz M, Matadamas-Hernandez N, Camacho-Casillas R, Magana-Magana R, Rojel-Martinez U, Alcocer-Gamba MA, Lara-Vaca S, Rodriguez-Reyes H, Islava-Galvez MA, Betancourt-Hernandez LE, Reyes-Reyes N, Beltran-Gamez ME, Cantu-Brito C, Banos-Velasco AZ, Del Rivero Morfin PJ, Gonzalez-Hermosillo JA. Anticoagulation Therapy by Age and Embolic Risk for Nonvalvular Atrial Fibrillation in Mexico, an Upper-Middle-Income Country: The CARMEN-AF Registry. Glob Heart. 2020 Apr 10;15(1):32. doi: 10.5334/gh.767. PMID 32489805